CLINICAL TRIAL: NCT04286737
Title: The Effect of Therapeutic Touch on Colic Symptoms in Infantile Colic Infants: A Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Selda Ateş Beşirik, Karamanoğlu Mehmetbey University, Faculty of Health Science, Pediatric Nursing Department, Karamanoğlu Mehmetbey University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019/2123
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Infantile Colic; Therapeutic Touch
Keywords: Therapeutic Touch; infantile colic; infant; nursing; Symptom
MeSH Terms: conditions — Colic | interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: The study will be conducted as a single-blind, randomized controlled trial.
Who Masked: Participant
Masking Description: Single blind will be done in the study. Only parents will be blinded. Two weeks follow up will be done in both groups. Since the researcher should implement the intervention, evaluate and manage the process, it will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Therapeutic Touch will be applied to infants for 3 consecutive days, once a day, 10 minutes at any time during the day. There will be a four-day break. The Therapeutic Touch will be done a total of 6 times in 2 weeks.
  Interventions: Other: Therapeutic Touch
- Control Group (No Intervention): The therapeutic touch will not be applied to the control group infants. However, the routine follow-up and behavior of the weekly baby will be evaluated to ensure that parents are blind.

INTERVENTIONS:
Other: Therapeutic Touch — Therapeutic Touch will be applied to infants for 3 consecutive days, once a day, 10 minutes at any time during the day. There will be a four-day break. The Therapeutic Touch will be done a total of 6 times in 2 weeks.
  Arms: Intervention Group

SUMMARY:
Aim: The purpose of this study is to determine the effect of therapeutic touch applied to infants with infantile colic on infant colic scale score, crying and sleep time.

Method: The study will be conducted as a single-blind, randomized controlled trial. The population of the study will be infants who come to the Pediatrics Outpatient Clinic and are diagnosed as infantile colic according to the evaluation of the pediatrician and have no other health problems. The infants will be divided into two groups as intervention and control groups according to stratified block randomization in the computer environment. After the randomization, therapeutic touch will be applied to the intervention group. No method will be applied to the control group.

DETAILED DESCRIPTION:
The research will be carried out with two groups as intervention and control groups. Sample size of the study has been determined by the power analysis, in line with the results obtained from the studies which have been conducted using a similar research method. According to the analysis results, it has been calculated as 27 for each group and 54 in total. Considering the possible case losses, 20% of the sample was increased. The sample consisted of 64 babies, 32 intervention and 32 control. Mothers of the infants meeting the study inclusion criteria will be informed both in written and verbally. Written consent will be obtained. The infants will be divided into two groups according to stratified block randomization in the computer environment. The infants will be stratified by gender and age. After the randomization, therapeutic touch will be applied to the intervention group. No method will be applied to the control group by the researcher. In obtaining research data, 4 tools will be used: "Mother-infant Information Form", "Infantile Colic Scale", Crying Time Registration Form and Sleep Time Registration Form.

ELIGIBILITY:
Inclusion Criteria:

* Family volunteering to participate in the research
* The infant was born at term
* The infant is between 4 weeks and 12 weeks
* The birth weight is between 2500-4500 g
* The infant has been diagnosed with infantile colic according to Wessel criteria
* Mothers' ability to read, write and speak Turkish
* New diagnosis of infantile colic

Exclusion Criteria:

* The infant has any chronic illness and congenital anomaly
* Mothers have diagnosed mental and mental problems
* Mother smoking
* The diagnosis of lactose intolerance to infants by the physician

Ages: 4 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-10-11 (Actual)

PRIMARY OUTCOMES:
Infantile Colic Scale | In two weeks
  Ellet et al. (2002) developed a Likert-type scale to determine the factors causing colic and to diagnose colic. Cetinkaya and Başbakkal (2007) tested the validity and reliability of the scale for the Turkish population. The scale consists of 5 sub-dimensions and 19 items.The low total score average from the scale indicates that the colic decreases, and the high average score indicates that the colic increases.

SECONDARY OUTCOMES:
Crying Time | In two weeks
  Infants' weekly crying times will be recorded.
Sleeping Time | In two weeks
  Infants' weekly sleeping times will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Selda Ateş Beşirik, Res. Assist., Principal Investigator — Karamanoğlu Mehmetbey University; Emine Geçkil, Professor, Study Director — Necmettin Erbakan University
Locations (1):
- Karaman Education and Research Hospital, Karaman, Turkey (Türkiye)